CLINICAL TRIAL: NCT02697565
Title: Healthy Caregivers-Healthy Children (HC2) Phase II: Integrating Culturally Sensitive Childhood Obesity Prevention Strategies Into Policy
Brief Title: Healthy Caregivers-Healthy Children (HC2) Phase II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Ruby Natale, Associate Professor of Clinical Pediatrics, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20140876; 2015-68001-23232 (Other Grant/Funding Number: USDA)
Record Dates: First submitted 2015-12-21; First posted 2016-03-03 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Pediatric Obesity; Obesity
Keywords: childhood obesity; obesity; prevention; nutrition; health; preschool; childcare; role model; pediatric obesity; weight; overweight; early childhood; train the trainer
MeSH Terms: conditions — Pediatric Obesity; Obesity; Body Weight; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Train-the-Trainers Arm (Experimental): Intervention Arm receives the Healthy Caregivers- Healthy Children Toolkit (healthy lifestyle role modeling intervention) via a nutritional gate keeper. The toolkit reinforces center health and activity policy standards.
  Interventions: Behavioral: Healthy Caregivers- Healthy Children Toolkit
- Attention Control Arm (Other): Control Arm that receives an attention control safety curriculum.
  Interventions: Behavioral: Safety Curriculum

INTERVENTIONS:
Behavioral: Healthy Caregivers- Healthy Children Toolkit — The treatment arm will receive the train-the-trainer model (utilizing Quality Counts coaches) to deliver the evidence- based HC2 toolkit.
  Arms: Train-the-Trainers Arm
Behavioral: Safety Curriculum — Centers randomized to the control arm will receive an attention control consisting of three visits from 'Safety Sam,' a character and safety curriculum that was fully developed and implemented in phase I of HC2. The same delivery model (train-the-trainers utilizing Quality Counts coaches) will be implemented.
  Arms: Attention Control Arm

SUMMARY:
One in four U.S. children under the age of 5 years old are either overweight or obese with ethnic-minority children being disproportionately affected. Low-income preschool children, many from ethnic minority backgrounds, receive childcare in federal/state subsidized centers where daily meals are provided. Nationally, the Quality Rating and Improvement Systems (QRIS) organization is responsible for rating the quality of childcare centers. However, nutrition and physical activity policy standards have not been incorporated into QRIS childcare center policies. Therefore, the goal of this project is to address the 2014 AFRI program area priority of Childhood Obesity Prevention by building on the phase I "Healthy Caregivers, Healthy Children (HC2)" NRI/AFRI funded project (2010-2013), in partnership with the Miami Dade County Cooperative Extension team, to evaluate the program via randomized-controlled trial outcomes, and deliver an evidence-based effective childcare center-based program/toolkit. This project (phase II) will expand HC2 Phase I findings by transferring the evidence-based HC2 program/toolkit to QRIS childcare centers via a train-the-trainers (TTT) model. The following specific aims are proposed; (1) to evaluate the TTT model of delivery for the evidence-based HC2 toolkit's effectiveness versus an attention control on parent and teacher adoption of healthy lifestyle role modeling behaviors, and policy integration; (2) to evaluate the impact of a TTT delivery model versus an attention control on child body composition and short- and long-term behavioral health outcomes, and (3) to disseminate the HC2 early childhood obesity prevention toolkit TTT model within the QRIS early childhood network at the Miami Dade County-level.

DETAILED DESCRIPTION:
While all states are responsible for childcare licensing standards, 26 states serving over 1 million preschool-age children currently implement QRIS. In MDC, QRIS-affiliated childcare facilities (collectively called Quality Counts or QC centers from this point forward) provide care to 1/3 of MDC's preschool-age children (80% are ethnic minorities) in 417 centers. At this time there are no nutrition policies included in the QRIS standards for childcare centers. Therefore, in light of the current childhood obesity epidemic, this project will address a major gap in knowledge and the disparities in access to healthy food consumption in the childcare center setting through HC2 implementation.

This study builds on previously funded work and will maximize the initial 3-year (2010-2013) investment the USDA made in phase I of the project to test effective obesity prevention strategies in the early childhood setting utilizing both educators and parents as nutritional gatekeeper, healthy lifestyle role models for 2-to-5 year-old children. The goal of this proposed project (phase II) is to expand the phase I evidence-based HC2 findings by giving ownership of the program/toolkit to the childcare centers via a train-the-trainers model and by implementing nutrition and physical activity standards into the Quality Rating Improvement System.

The proposed integrated project is responsive to the USDA's National Institute of Food and Agriculture (formerly CSREES) functions by addressing all three areas of the agricultural knowledge system, including (1) a scientifically-based and rigorous Research design that assesses obesity prevention efforts with young children in a novel setting of childcare facilities; (2) the development of an Educational tool kit to improve training and capacity of teachers and parents/families. Extension and capacity building will be enhanced through HC2 toolkits delivered to the centers and train-the-trainer program manuals for use throughout the QRIS network and in cooperation with Florida FNP. Finally, by incorporating HC2 practices into permanent QRIS policy, centers can sustain the project's benefits for future children, teachers, and families. Additionally, the investigators will collaborate with two community nutritionists to provide services to a large number of childcare centers in the county therefore, extending project materials. Lastly, the toolkit will sustain education and extension functions beyond the life of the project by giving ownership of HC2 to the childcare centers.

ELIGIBILITY:
Inclusion Criteria:

* QC centers must meet the following criteria to be included: (1) have > 30 children ages 2-5 enrolled; (2) Serve low income families; (3) be a part of the USDA food program and Supplemental Nutrition Assistance Program (SNAP) eligible; (3) Reflect the ethnic diversity of the MDC Public School System (63 percent Hispanic, 19 percent African American, 18 percent white); and (4) Center directors agree to participate and sign a letter of commitment (see Documents of Collaboration).

Exclusion Criteria:

* Centers with a high prevalence of special needs children.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2289 (Actual)
Dates: Start 2015-04; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Change in The Environment and Policy Assessment and Observation tool (EPAO) score | 3 years
  The EPAO will examine childcare center environmental changes. The EPAO will assess the level of implementation of the snack, screen time, physical activity, and beverage policies through direct observation of diet and physical activity. Child health behaviors and parent and teacher health behaviors will also be measured.

SECONDARY OUTCOMES:
Observed pre-post maintenance on Child's Body Mass Index (BMI) | 2 years
  BMI is based on height and weight of the child as per CDC guidelines
Change of caregiver role modeling behavior | 2 years
  The HC2 self assessment tool has a role modeling scale, measuring role modeling behavior

CONTACTS AND LOCATIONS:
Overall Officials: Ruby Natale, PhD, PsyD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

REFERENCES:
- [Background] Messiah SE, Arheart KL, Natale RA, Hlaing WM, Lipshultz SE, Miller TL. BMI, waist circumference, and selected cardiovascular disease risk factors among preschool-age children. Obesity (Silver Spring). 2012 Sep;20(9):1942-9. doi: 10.1038/oby.2011.353. Epub 2011 Dec 8. PMID 22158004
- [Background] Natale R, Scott SH, Messiah SE, Schrack MM, Uhlhorn SB, Delamater A. Design and methods for evaluating an early childhood obesity prevention program in the childcare center setting. BMC Public Health. 2013 Jan 28;13:78. doi: 10.1186/1471-2458-13-78. PMID 23356862
- [Background] Natale R, Page M, Sanders L. Nutrition and physical activity practices in childcare centers versus family childcare homes. Early Childhood Educ J. 2013; [Epub] DOI 10.1007/s10643-013-0607-4.
- [Background] Natale RA, Messiah SE, Asfour L, Uhlhorn SB, Delamater A, Arheart KL. Role modeling as an early childhood obesity prevention strategy: effect of parents and teachers on preschool children's healthy lifestyle habits. J Dev Behav Pediatr. 2014 Jul-Aug;35(6):378-87. doi: 10.1097/DBP.0000000000000074. PMID 25007060
- [Background] American Academy Of Pediatrics, American Public Health Association, National Resource Center for Health and Safety in Child Care and Early Education. 2011. Caring for our Children: National health and safety performance standards; Guidelines for early care and education programs. 3rd edition. Elk Grove Village, IL: American Academy of Pediatrics; Washington, DC: American Public Health Association. Available at http://nrckids.org.
- [Background] McGuire S. Institute of Medicine (IOM) Early Childhood Obesity Prevention Policies. Washington, DC: The National Academies Press; 2011. Adv Nutr. 2012 Jan;3(1):56-7. doi: 10.3945/an.111.001347. Epub 2012 Jan 5. No abstract available. PMID 22332102
- [Background] Derananian CA, Desai P, Smith-Ray R, Seymour RB, Hughes SL. Perceived versus actual factors associated with adoption and maintenance of an evidence-based physical activity program. Transl Behav Med. 2012 Jun;2(2):209-17. doi: 10.1007/s13142-012-0131-x. PMID 24073112
- [Background] Ball SC, Benjamin SE, Hales DP, Marks J, McWilliams, P, Ward DS. The Environment and Policy Assessment and Observation (EPAO) Child Care Nutrition and Physical Activity Instrument. Chapel Hill, NC: Center for Health Promotion and Disease Prevention, University of North Carolina at Chapel Hill; 2005.
- [Background] Ball SC, Benjamin SE, Ward DS. Development and reliability of an observation method to assess food intake of young children in child care. J Am Diet Assoc. 2007 Apr;107(4):656-61. doi: 10.1016/j.jada.2007.01.003. PMID 17383271
- [Background] Benjamin SE. Preventing Obesity in the Child Care Setting: Evaluating State Regulations. http://cfm.mc.duke.edu/wysiwyg/downloads/State_Report-NC.pdf. Accessed October 22, 2010.
- [Background] Benjamin SE, Ammerman A, Sommers J, Dodds J, Neelon B, Ward DS. Nutrition and physical activity self-assessment for child care (NAP SACC): results from a pilot intervention. J Nutr Educ Behav. 2007 May-Jun;39(3):142-9. doi: 10.1016/j.jneb.2006.08.027. PMID 17493564
- [Background] Townsend MS, Slyva K, Davidson C, Leavens L, Sitnick SL, Design: Chao LK. Healthy Kids: Pediatric Obesity Risk Assessment Tool. [45 items reflecting 23 behaviors and 12 determinants of obesity identified in our research.] University of California Cooperative
- [Background] McAlearney, Edwards. Organizational Readiness to Change Survey, Version 2.0. Published 2008. http://www.rwjf.org/content/dam/files/rwjf-web-files/Resources/1/esorganizationalreadinesssurvey.pdf. Accessed January 12, 2014.
- [Background] Willett WC, Sampson L, Stampfer MJ, Rosner B, Bain C, Witschi J, Hennekens CH, Speizer FE. Reproducibility and validity of a semiquantitative food frequency questionnaire. Am J Epidemiol. 1985 Jul;122(1):51-65. doi: 10.1093/oxfordjournals.aje.a114086. PMID 4014201
- [Background] Townsend M, Kaiser L, Graphic Designer: Chao LK. Fruit and Vegetable Inventory. http://townsendlab.ucdavis.edu/PDF_files/FV/FV_Inventory.pdf. Accessed March 25, 2014.
- [Background] Marcus BH, Selby VC, Niaura RS, Rossi JS. Self-efficacy and the stages of exercise behavior change. Res Q Exerc Sport. 1992 Mar;63(1):60-6. doi: 10.1080/02701367.1992.10607557. PMID 1574662
- [Background] Parcel GS, Edmundson E, Perry CL, Feldman HA, O'Hara-Tompkins N, Nader PR, Johnson CC, Stone EJ. Measurement of self-efficacy for diet-related behaviors among elementary school children. J Sch Health. 1995 Jan;65(1):23-7. doi: 10.1111/j.1746-1561.1995.tb03335.x. PMID 7731197
- [Background] U.S. Department of Health and Human Services, HRSA: Health Resources and Services. Growth Charts Training. Administration, Maternal and Child Health Bureau,. Hyattsville, MD: U.S. Department of Health and Human Services, Centers for Disease Control and Prevention; 2008. http://www.cdc.gov/NCHS/data/nhanes/ nhanes_01_02/body_measures_year_3.pdf. Accessed January 5, 2014.
- [Background] Messiah SE, Arheart KL, Luke B, Lipshultz SE, Miller TL. Relationship between body mass index and metabolic syndrome risk factors among US 8- to 14-year-olds, 1999 to 2002. J Pediatr. 2008 Aug;153(2):215-21. doi: 10.1016/j.jpeds.2008.03.002. Epub 2008 Apr 18. PMID 18534237
- [Background] Ogden CL, Carroll MD, Kit BK, Flegal KM. Prevalence of obesity and trends in body mass index among US children and adolescents, 1999-2010. JAMA. 2012 Feb 1;307(5):483-90. doi: 10.1001/jama.2012.40. Epub 2012 Jan 17. PMID 22253364
- [Background] Nader PR, O'Brien M, Houts R, Bradley R, Belsky J, Crosnoe R, Friedman S, Mei Z, Susman EJ; National Institute of Child Health and Human Development Early Child Care Research Network. Identifying risk for obesity in early childhood. Pediatrics. 2006 Sep;118(3):e594-601. doi: 10.1542/peds.2005-2801. PMID 16950951
- [Background] U.S. Center for Disease Control, National Center for Chronic Disease Prevention and Health Promotion, Division of Nutrition, Physical Activity and Obesity. Obesity among low-income preschool children. Retrieved June 16, 2014 from http://www.cdc.gov/obesity/downloads-/PedNSSFactSheet.pdf
- [Background] Birch LL, Anzman SL. Learning to eat in an obesogenic environment: A developmental systems perspective on childhood obesity. Child Dev Persp. 2010; 4:138-143.
- [Background] Ogden CL, Carroll MD, Flegal KM. High body mass index for age among US children and adolescents, 2003-2006. JAMA. 2008 May 28;299(20):2401-5. doi: 10.1001/jama.299.20.2401. PMID 18505949
- [Background] Everson-Hock ES, Johnson M, Jones R, Woods HB, Goyder E, Payne N, Chilcott J. Community-based dietary and physical activity interventions in low socioeconomic groups in the UK: a mixed methods systematic review. Prev Med. 2013 May;56(5):265-72. doi: 10.1016/j.ypmed.2013.02.023. Epub 2013 Feb 27. PMID 23454537
- [Background] Natale R, Messiah SE, Lopez-Mitnik G, Barth J, Sanders L. Prevalence of overweight and related health behaviors in an inner-city minority preschool population. Int J Interdisc Soc Sci. 2008;(3)4:17-28.
- [Background] Fox M, Glantz F, Endahl J, J. W. Early Childhood and Child Care Study. Alexandria, VA: 1 Bibliography & References Cited U.S. Department of Agriculture; 1997.
- [Background] Fitzgibbon ML, Stolley MR, Dyer AR, VanHorn L, KauferChristoffel K. A community-based obesity prevention program for minority children: rationale and study design for Hip-Hop to Health Jr. Prev Med. 2002 Feb;34(2):289-97. doi: 10.1006/pmed.2001.0977. PMID 11817926
- [Background] Zenk SN, Schulz AJ, Israel BA, James SA, Bao S, Wilson ML. Neighborhood racial composition, neighborhood poverty, and the spatial accessibility of supermarkets in metropolitan Detroit. Am J Public Health. 2005 Apr;95(4):660-7. doi: 10.2105/AJPH.2004.042150. PMID 15798127
- [Background] Glasgow RE, Vogt TM, Boles SM. Evaluating the public health impact of health promotion interventions: the RE-AIM framework. Am J Public Health. 1999 Sep;89(9):1322-7. doi: 10.2105/ajph.89.9.1322. PMID 10474547
- [Background] McGarvey E, Keller A, Forrester M, Williams E, Seward D, Suttle DE. Feasibility and benefits of a parent-focused preschool child obesity intervention. Am J Public Health. 2004 Sep;94(9):1490-5. doi: 10.2105/ajph.94.9.1490. PMID 15333300
- [Background] Bandura A. Social Foundations of Thought and Action: A Social Cognitive Theory. Upper Saddle River, NJ: Prentice Hall;1986.
- [Derived] Messiah SE, Lebron C, Moise R, Sunil Mathew M, Sardinas K, Chang C, Palenzuela J, Walsh J, Shelnutt KP, Spector R, Altare F, Natale R. Healthy caregivers-healthy children (HC2) phase 2: Integrating culturally sensitive childhood obesity prevention strategies into childcare center policies. Contemp Clin Trials. 2017 Feb;53:60-67. doi: 10.1016/j.cct.2016.12.011. Epub 2016 Dec 12. PMID 27979753